CLINICAL TRIAL: NCT00229749
Title: Exploratory Study of AVI-4065 Injection to Design Therapeutic Dosing for Chronic Active HCV Patients
Brief Title: Study of AVI-4065 in Healthy Volunteers and Chronic Active HCV Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Limited viral load reduction in HCV subjects
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4065-20
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: AVI-4065 Injection

SUMMARY:
Chronic active hepatitis C viral infections are difficult to treat: current drug therapies can result in severe side effects that some patients will not tolerate. AVI-4065 Injection is a new drug designed to prevent the virus from reproducing in the body. We tested this drug in healthy adult volunteers to optimize the dosing regimen, and are now proceeding in adult patients with chronic active hepatitis C infections. Patients who have the disease and who have had treatment but without success, will be recruited for the study.

The treatment of HCV patients initially consisted of subcutaneous injections given twice a day for 14-days. Treatment arms of 28 days, twice or three-times per day have been added.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is the most common blood-borne infection in the United States and a worldwide public health problem of epidemic proportions. Benign in the acute phase of infection, HCV infection usually becomes chronic in 70% of those originally infected. Chronic HCV infection leads to inflammation of the liver (hepatitis), cirrhosis, end-stage liver disease, and hepatocellular carcinoma. In the United States alone, there are over 2.7 million individuals with chronic HCV hepatitis. Standard treatment of chronic HCV hepatitis is combination therapy for 24 to 48 weeks with alpha interferon and ribavirin. This combination has limited efficacy, poor tolerability, and significant expense in terms of drug and ancillary laboratory testing. It is well recognized that new treatment options are needed which are more efficacious, potent, less toxic, and less expensive.

AVI BioPharma has pursued discovery of a drug against HCV using proprietary Neugene® or Phosphorodiamidate Morpholino Oligomer (PMO) synthetic chemistry. Neugene (PMO) compounds, as a drug class, are considered safe in humans and do not activate complement, alter clotting times, or bind to α-adrenergic receptors (which can produce hypotension) like the phosphorothioate antisense compounds. One PMO, AVI-4065, has been identified as likely to inhibit all 5 genotypes of HCV based on in vitro and in vivo animal models. There are specific data that confirm that AVI-4065 can inhibit HCV RNA dependent PNA polymerase (RdRp encoded in NS5) and the HCV protease (NS3), in a non-competitive inhibitory fashion. The 50 percent Effective Concentration (EC50) is 308 nM, and the efficacy is nearly 100% at 3 μM. These data suggest that AVI-4065 is capable of inhibiting HCV protein translation in a robust manner at concentrations that should be achievable in patients. In rigorous GLP safety pharmacology and toxicity models in a variety of animal species at dosage levels up to 5 times the maximum anticipated human dosage level, inclusive of non-human primates, AVI-4065 was considered safe, well tolerated and without dose-limiting toxicities. Additionally, AVI-4065 Injection was safe and well-tolerated in the three dose-escalating groups of 31 healthy volunteers (Part I) with no serious adverse events. Adverse events that did occur were few, self-limited and mild to moderate and did not require intervention; this observation held true for the first HCV patients receiving AVI-4065 Injection.

AVI BioPharma's first human use of AVI-4065 Injection involved an open-label, multi-center, exploratory, dose escalating design in healthy adult volunteers. The objective of this part of the study was to assess safety, tolerability and to design a potentially therapeutic dosage regimen. The objective of the second part of the study is to evaluate safety, tolerability, pharmacokinetics, pharmacodynamics and signals of HCV virus response in cohorts of HCV patient volunteers that are interferon and ribavirin treatment failures.

The ability of the drug to effect baseline HCV RNA levels over the study duration will be evaluated using a conventional PCR-based assay. If there are promising results from this phase of the clinical trial (viz., a 2 log decrease in HCV RNA levels from baseline within study surveillance), it will provide the rational basis for additional clinical testing of AVI-4065 Injection among HCV patients that are treatment refractory (viz., relapsers and non-responders).

ELIGIBILITY:
Inclusion Criteria - Part II: (HCV Infected Patients)

* Adult males and females aged 18 to 64 years of age
* Chronic HCV infection, defined as virological diagnosis of HCV for at least six months with detectable serum HCV-RNA levels >100,000 IU/mL by an HCV-RNA PCR assay on two occasions at least one week apart within 4 weeks prior to study drug administration
* Signed and dated written informed consent form
* Negative serum ß-HCG (pregnancy) test 24 hours prior to initial dose of AVI-4065 Injection for females of childbearing potential, or post-menopausal and amenorrheic for 2 years, or surgically sterilized for at least one year
* Willing to abstain from alcohol from the beginning of study entry through Day 28 of the study
* Willing to participate in all study activities (including the ability to safely self-inject study drug subcutaneously) and all study requirements (including effective contraception) during study period

Exclusion Criteria - Part II (HCV Patients):

* Hematology, coagulation, serum chemistry, and urinalysis laboratory test values >2 times upper limits of normal or anemia (hemoglobulin <11 g/dL), leukopenia (total white blood count <3,000/ µL or total neutrophils <1,500/ µL) or thrombocytopenia (platelets <100,000/ µL)
* Decompensated or severe liver disease, defined as cirrhotic patients with a Child-Pugh score of ≥ 7
* Encephalopathy or altered mental status of any etiology
* Any neoplasm, including hepatocellular carcinoma
* Decompensated renal disease (e.g., serum creatinine >2.5 or on a dialysis program)
* Positive HIV-1 or HIV-2 serology
* Positive Hepatitis B Surface Antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb) status
* Participation in any interventional clinical trial within previous 6 months
* Organ transplant recipient (solid or hematopoietic)
* Use of interferons and ribavirin or experimental HCV treatment within past 6 months
* Use of non-steroidal anti-inflammatory agents (e.g., ibuprofen, naproxen or COX-2 inhibitors) that exceeds 2 days per week of the recommended daily dosing or usage that exceeds 5 grams/week.
* Use of acetaminophen within 15 days of enrollment and throughout Day 28 of the study
* Body Mass Index (BMI) > 35
* Pregnant or nursing female
* Active serious or poorly controlled chronic illness
* History of poor compliance with health and treatment regimens
* Use of herbal or homeopathic products, illicit drugs, statins, corticosteroids, immunosuppressives, or cytotoxic agents within 90 days of first dose of study drug
* Use of drugs with potential hepatotoxicity, e.g., oral antifungals or oral glucophage inhibitors
* Unwilling to participate in any study activity (including to safely self-inject study medication subcutaneously) and complete any study requirement (including effective contraception) during study period and competition of any study visit
* Investigator opinion of unsuitability

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability
Pharmacokinetics/pharmacodynamics

SECONDARY OUTCOMES:
Response of HCV levels to AVI-4065 Injection, via serum HCV-RNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Mark Holodniy, M.D., Principal Investigator — Stanford University School of Medicine and Department of Veterans Affairs Public Health Research & Consultation Program at the Veterans Affairs Palo Alto Health Care System